CLINICAL TRIAL: NCT01587599
Title: Pharmaceutical Care of Elderly Diabetes-patients With Impaired Mobility in a Model-region of Decreasing Supply of Medical Services in North-eastern Germany
Brief Title: Pharmaceutical Care of Patients With Impaired Mobility in a Model-region of Decreasing Supply of Medical Services
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foerderinitiative Pharmazeutische Betreuung e.V. (Other)
Responsible Party: Principal Investigator, Prof. Dr. Christoph Ritter, Professor of Clinical Pharmacy, Foerderinitiative Pharmazeutische Betreuung e.V.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FI_CLIN_PHARM_EMAU_01
Record Dates: First submitted 2012-04-25; First posted 2012-04-30 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes
Keywords: pharmaceutical care; drug-related problems; elderly; Pharmaceutical care of elderly patients with diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmaceutical care (Active Comparator)
  Interventions: Behavioral: counseling
- Standard care (Placebo Comparator)
  Interventions: Behavioral: counseling

INTERVENTIONS:
Behavioral: counseling — The patients grouped to the intervention cohort receive pharmaceutical care by a pharmacist during the study period.

SUMMARY:
Design and Procedure:

The design is a randomised controlled multi-centre pilot study. 18 community pharmacies located in Mecklenburg-Western Pomerania, Germany, were randomised to either a control or an intervention group. These pharmacies recruited eligible patients out of their clientele and invited them to take part in the study. Participants were visited at home by the pharmacist and home-based medication reviews were conducted. The survey form has been developed by the research team and comprised amongst others items to adherence, adverse effects, drug intake, storage and quality of life. Thereafter all data were analysed by the pharmacist with a newly developed document called "analysis guide" aiming at the detection of drug related problems. Pharmacists of the intervention group discussed the results with the family doctor of the patients and the patients and tried to solve the drug related problems. This procedure was not undertaken in the control group.

Six months later a second medication review was carried out in both groups.

Study hypothesis:

Pharmaceutical care reduces the overall number of drug-related problems of elderly patients with diabetes and impairments in mobility.

Aim:

The purpose of this study is to show that pharmaceutical care reduces the overall number of drug-related problems of elderly diabetes-patients with impairments in mobility and leads to both an improved health status and an improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* impairment in mobility
* age of 65 years or older
* four or more long-term medications
* diabetes
* at least one of the following co-morbidities: hypertension, obesity, hypercholesteremia, hyperlipidemia, coronary heart disease, cardiac insufficiency, angina pectoris, peripheral vascular disease

Exclusion Criteria:

* patient lives in a home for the aged or a residential care home for the elderly
* terminal renal failure, dialysis
* moderately or severe dementia or other severe cognitive impairments
* terminal diseases (e.g. cancer)
* nursing service if the medicine is directly administered to the patient

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
adherence | 6 months
  MMAS-8d
adverse events | 6 months
  SHIP-trend 8-items questionnaire
drug-drug-interactions | 6 months
  ABDATA drug-drug interaction identification tool

SECONDARY OUTCOMES:
quality of life | 6 months
  improvement of quality of life, measured with eq-5d
improved overall health status | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A Ritter, Prof. Dr., Principal Investigator — Ernst-Moritz-Arndt-University Greifswald, Germany